CLINICAL TRIAL: NCT01831453
Title: Therapeutic Effect of Systemic Omega-3 Polyunsaturated Fatty Acids On Quality of Life in Patients Suffering From Recurrent Aphthous Stomatitis Unresponsive to Topical Therapy.
Brief Title: Omega-3 and Quality of Life in Recurrent Aphthous Stomatitis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Moustafa Elkhouli, Associate professor, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr. Amr Elkhouli 1962
Record Dates: First submitted 2013-04-05; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Mouth Ulcers
Keywords: omega-3; recurrent aphthous stomatitis; quality of life
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Docosahexaenoic Acids; Fish Oils; isopropyl myristate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- isopropylmyristate oil (Placebo Comparator): placebo Soft gelatinous capsules filled with isopropylmyristate oil
  Interventions: Drug: placebo
- experimental (Active Comparator): omega-3 1 gram three times daily for 6 months
  Interventions: Drug: omega-3

INTERVENTIONS:
Drug: omega-3 — polyunsaturated fatty acids(PUFAs) 1 gram three times per day for 6 months
  Other Names: fish oil
  Arms: experimental
Drug: placebo — soft gelatinous capsules filled with isopropylmyristate oil
  Other Names: isopropylmyristate oil
  Arms: isopropylmyristate oil

SUMMARY:
The study aims at evaluating the effect of omega-3 on patients suffering recurrent oral aphthous ulcers

DETAILED DESCRIPTION:
In this study, we tested the hypothesis that the administration of omega 3 improve the quality of life in patients suffering recurrent oral ulceration and improve associated symptoms of pain in addition to reduction of ulcers episode.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients older than 13 years of age
2. Presenting with 1 to 3 aphthous ulcers (less than 48 hours' duration) with a size no greater than 5mm in diameter.
3. History of recurrent minor aphthous ulcer for at least one year with a frequency of at least one outbreak every one month.
4. Normal sense of pain, without anesthesia or paresthesia.
5. Willingness to participate and sign the informed consent.

Exclusion Criteria:

* 1- Concurrent clinical conditions that could pose a health risk to the subjects including serious heart, liver, or kidney dysfunctions.

  2- Pregnancy and lactation. 3- Ulcers as a manifestation of systemic disorders such as Ulcerative Colitis, Crohn's disease, Behçet's syndrome or serious anemia.

  4- Treatment with systemic steroids, immunomodulatory agents, antibiotics, non-steroidal anti-inflammatory drugs (except occasional use for headaches) one month prior to the study entry.

  5- Treatment of the current ulcer with any topical or systemic medication. 6- Attendance of any other clinical trials prior to 3 months of study entry.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
quality of life | six months
  Measurement of oral health related quality of life (OHR-QoL),this parameter was carried out at baseline, and at 6 months of the study using the Arabic version of oral health impact profile-14 (OHIP-14) questionnaire.

SECONDARY OUTCOMES:
Pain associated with the ulcers | Six months
  The measurements for treatment effectiveness included evaluation of pain associated with the ulcer(s) by means of visual analogue scales (VAS).
Duration of ulcers episode | Six months
  The time needed for the ulcer to heal
The monthly number of ulcer outbreaks | Monthly for six months
  The number of ulcers appears monthly in the mouth

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Elkhouli, ass prof, Principal Investigator — October 6 University
Locations (1):
- October 6 university, Cairo, Governarate of 6 of October, Egypt

REFERENCES:
- [Background] Hjorth E, Zhu M, Toro VC, Vedin I, Palmblad J, Cederholm T, Freund-Levi Y, Faxen-Irving G, Wahlund LO, Basun H, Eriksdotter M, Schultzberg M. Omega-3 fatty acids enhance phagocytosis of Alzheimer's disease-related amyloid-beta42 by human microglia and decrease inflammatory markers. J Alzheimers Dis. 2013;35(4):697-713. doi: 10.3233/JAD-130131. PMID 23481688
- See also: alzheimers — http://www.alzheimers.org/